CLINICAL TRIAL: NCT03802565
Title: Dose Ranging Study of Tolperisone in Acute Muscle Spasm of the Back
Brief Title: Tolperisone in Acute Muscle Spasm of the Back
Acronym: STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurana Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Back Pain; Acute Pain; Back Spasm Upper Back; Back Strain; Muscle Cramp; Muscle Spasm; Low Back Pain
MeSH Terms: conditions — Back Pain; Acute Pain; Muscle Cramp; Spasm; Low Back Pain | interventions — Tolperisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tolperisone 50 mg (Experimental): TID (150 mg/day)
  Interventions: Drug: Tolperisone
- Tolperisone 100 mg (Experimental): TID (300 mg/day)
  Interventions: Drug: Tolperisone
- Tolperisone 150 mg (Experimental): TID (450 mg/day)
  Interventions: Drug: Tolperisone
- Tolperisone 200 mg (Experimental): TID (600 mg/day)
  Interventions: Drug: Tolperisone
- Placebo (Placebo Comparator): TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolperisone — TID
  Arms: Tolperisone 100 mg; Tolperisone 150 mg; Tolperisone 200 mg; Tolperisone 50 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel group study of the efficacy and safety of tolperisone (a non-opioid) or placebo administered as multiple doses three times a day (TID) in approximately 400 male and female subjects experiencing back pain due to or associated with muscle spasm.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Current acute back pain and/or stiffness due to acute and painful muscle spasm starting within 7 days prior to study entry and more than 8 weeks after the last episode of acute back pain.
* Pain of 4 or more on the subject "right now" rating of pain intensity Numeric Rating Scale (NRS) scale of 0-10.
* Willing to discontinue all medication used for the treatment of pain or muscle spasm on study entry.
* Pain localized below the neck and above the inferior gluteal folds.
* Body mass index ranging between 18 and 35 kg/m².

Exclusion Criteria:

* Unwillingness to stop taking pain or antispasmodic medication other than the study medication (specifically opioid use [e.g., Vicodin], barbiturates, and cannabis).
* Chronic pain for the previous 3 months or longer, on more days than not.
* Radicular pain in the lower extremity (i.e. pain radiating below the knee), sciatica pain down the leg, or pain below the knee (indicating a lumber radiculopathy); radicular pain in the upper extremity, radiating into the forearm or hand (indicating a cervical radiculopathy).
* Concomitant severe pain in a region other than the back.
* Spinal surgery within 1 year of study entry.
* Back pain due to major trauma (e.g., motor vehicle accident, fracture of bone) unless resolved for more than 1 year.
* Treatment of back pain ongoing with non-pharmacological therapy (e.g., acupuncture, chiropractic adjustment, massage, Transcutaneous Electrical Nerve Stimulation [TENS], physiotherapy).
* Subjects who test positive for alcohol by breathalyzer test.
* Unwilling to stop taking moderate to potent inhibitors of cytochrome P450 (CYP) isozymes CYP2D6 and CYP2C19, which are likely to cause drug interactions with tolperisone HCl (e.g., medications such as paroxetine and fluvoxamine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Tennessee Valley Pain Consultants, Huntsville, Alabama
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Center of Applied Research, Little Rock, Arkansas
  - Research Center of Fresno, Fresno, California
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - Northern California Research, Sacramento, California
  - Pacific Research Network, LLC, San Diego, California
  - San Diego Sports Medicine, San Diego, California
  - CITrials, Santa Ana, California
  - Riverside Clinical Research, Edgewater, Florida
  - Empirical Research Group, Gainesville, Florida
  - LLC Medical Research, Miami, Florida
  - Savin Medical Group, Miami Lakes, Florida
  - Avail Clinical Research, Orange City, Florida
  - Private Practice, Plantation, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Georgia Clinical Research, Snellville, Georgia
  - MediSphere Medical Research Center, Evansville, Indiana
  - Otrimed Clinical Research, Edgewood, Kentucky
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Center for Rheumatology and Bone, Wheaton, Maryland
  - Michigan Head Pain and Neurological, Ann Arbor, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - Jubilee Clinical Research, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Upstate Clinical Research Associates, Williamsville, New York
  - Clinical Trials of America, Winston-Salem, North Carolina
  - Sterling Research Group- Springdale, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Center for Providence Health Partners, Dayton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Williamette Valley Clinical Studies, Eugene, Oregon
  - Frontier Clinical Research, Inc., Smithfield, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Inquest Clinical Research, Baytown, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - HD Research Corp, Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - ClinRX Research Joseph, Inc., Plano, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tolperisone 50 mg | Tolperisone 100 mg | Tolperisone 150 mg | Tolperisone 200 mg | Placebo
Started | 82 | 87 | 83 | 85 | 78
Completed | 77 | 83 | 74 | 77 | 72
Not Completed | 5 | 4 | 9 | 8 | 6
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 4 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Subjects Related to Each Other | 1 | 0 | 0 | 2 | 1
Not completed — Elevated Enzymes | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolperisone 50 mg | Tolperisone 100 mg | Tolperisone 150 mg | Tolperisone 200 mg | Placebo | Total
Number analyzed (Participants) | 82 | 87 | 83 | 85 | 78 | 415
Age, Customized [Mean (Full Range); unit: years] | 43.5 [20 to 65] | 44.4 [19 to 65] | 44.3 [21 to 65] | 42.0 [20 to 64] | 41.6 [18 to 62] | 43.6 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 57 | 41 | 41 | 49 | 233
  Male | 37 | 30 | 42 | 44 | 29 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 22 | 20 | 16 | 89
  Not Hispanic or Latino | 69 | 69 | 61 | 65 | 62 | 326
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 1 | 3
  Asian | 1 | 4 | 2 | 4 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 0 | 3
  Black or African American | 29 | 32 | 29 | 35 | 29 | 154
  White | 50 | 50 | 49 | 45 | 42 | 236
  More than one race | 0 | 0 | 1 | 0 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Body Mass Index [Mean (Full Range); unit: kilogram/meter^2] | 28.23 [19.4 to 35.0] | 28.48 [20.9 to 35.0] | 28.34 [19.8 to 35.0] | 28.45 [20.0 to 35.0] | 28.53 [19.5 to 35.0] | 28.38 [19.4 to 35.0]

OUTCOME MEASURES:

1. Primary Outcome: Mean Effect Size in Subjected-Rated Pain
Description: Mean effect size between Tolperisone and Placebo of subject-rated pain due to acute back spasm using a Numerical Rating Scale (NRS; 0-10 scale, from no pain to worst possible pain) on Day 14 "right now."
Time Frame: Day 1 to Day 14
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tolperisone 50 mg | Tolperisone 100 mg | Tolperisone 150 mg | Tolperisone 200 mg | Placebo
Number analyzed (Participants) | 82 | 87 | 83 | 85 | 78
score on a scale | -4.2 [-9 to 1] | -4.0 [-10 to 2] | -3.7 [-8 to 1] | -4.4 [-10 to 1] | -3.5 [-8 to 1]

ADVERSE EVENTS:
Time Frame: First Dose, Day 1 to Follow-up, Day 28
Arm/Group | Tolperisone 50 mg | Tolperisone 100 mg | Tolperisone 150 mg | Tolperisone 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/87 | 0/83 | 0/85 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/87 | 0/83 | 0/85 | 0/78
Other Adverse Events (participants affected / at risk) | 7/82 | 13/87 | 12/83 | 14/85 | 5/78
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolperisone 50 mg (N=82) | Tolperisone 100 mg (N=87) | Tolperisone 150 mg (N=83) | Tolperisone 200 mg (N=85) | Placebo (N=78)
Headache (Nervous system disorders) | 3 | 5 | 8 | 8 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03802565/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03802565/SAP_000.pdf